CLINICAL TRIAL: NCT01325844
Title: The Effects of Epidural Anesthesia on the Bioavailability of Nitric Oxide and Renal Function in Patients Undergoing Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2010-0537
Record Dates: First submitted 2011-03-28; First posted 2011-03-30 (Estimated); Last update posted 2012-02-06 (Estimated); Status verified 2012-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Anesthesia, Epidural

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- G group (No Intervention): G group = General anesthesia group
- G+E group (Experimental): G+E group = General anesthesia + epidural anesthesia group
  Interventions: Procedure: Epidural anesthesia

INTERVENTIONS:
Procedure: Epidural anesthesia — 0.5% ropivacaine infusion via epidural catheter at 5ml/hr during general anesthesia
  Arms: G+E group

SUMMARY:
This study was designed to investigate the effects of epidural anesthesia combined with general anesthesia during laparoscopic surgery. The investigators hypothesized that epidural anesthesia will effectively block the activation of the sympathetic nervous system during surgery, thus activating nitric oxide and reducing splanchnic ischemia and decrease in postoperative renal function.

ELIGIBILITY:
Inclusion Criteria:

* ASA class 1 or 2 adult patients scheduled for endoscopic prostatectomy

Exclusion Criteria:

* Patient refusal
* Patients on diuretics
* Patients with renal failure (eGFR < 60 ml/min/1.73 m2)

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-11; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
blood pressure with heart rate variability | 10 minutes after anesthesia induction

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea